CLINICAL TRIAL: NCT04602897
Title: The Analgesic Efficacy of Forced Coughing During Intrauterine Device Insertion: A Randomized Clinical Trial
Brief Title: The Analgesic Efficacy of Forced Coughing During Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Nabih Elkhouly, Asssistant professor of obstetrics and gynecology, Menoufia University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-2019OBSGN38
Record Dates: First submitted 2020-10-16; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Pain
Keywords: Intrauterine device, IUD, Pain, Forced coughing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The cough group patients were asked to cough a forced cough during different steps of IUD insertion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cough group (Experimental): The cough group patients were asked to cough a forced cough during different steps of IUD insertion
  Interventions: Other: forced coughing
- control (No Intervention): the control group received no pain management at all during different steps of IUD insertion

INTERVENTIONS:
Other: forced coughing — The cough group patients were asked to cough a forced cough during different steps of IUD insertion
  Arms: cough group

SUMMARY:
This was a randomized controlled trial of 400 women who attended the outpatient clinic of Menoufia University Hospital for copper IUD insertion. The women were randomly assigned to cough and control groups.The primary outcome measure was the level of pain experienced at different steps of IUD insertion measured by a visual analogue scale (VAS).

DETAILED DESCRIPTION:
We conducted this randomized controlled trial at the Department of Obstetrics and Gynecology at Menoufia University Hospital, Egypt, from May 2018 to March 2020. Our hospital research ethics committee approved this study. We obtained informed consent from all participants before initiating any study procedures. CONSORT guidelines were observed and completed.

We recruited non pregnant women (aged 18-45 years) requesting copper T380A IUD insertion for contraception. Eligible women had no prior vaginal delivery or pregnancy termination beyond 12 weeks, gestation (as patulous cervical os may affect VAS score), any previous deliveries had been by cesarean section, they were immediately postmenstrual or 1 week after pregnancy termination and they were willing to complete the study questionnaires. All women had to be alert, oriented, and cooperative to respond easily to VAS.

Exclusion criteria were current pregnancy, prior vaginal delivery, history of cervical stenosis, current pelvic inflammatory disease, uterine anomalies, undiagnosed abnormal uterine bleeding, fibroids distorting the uterine cavity, and patients using chronic NSAIDs or on chronic pain medication.

We randomized participants in a 1:1 ratio to cough and control groups. A statistician not directly involved in the study prepared a computer generated randomization list and placed the allocation information in sequentially numbered sealed envelopes that were opened according to the attendance of the subjects after signing the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant women (aged 18-45 years) requesting copper T380A IUD insertion for contraception.
* No prior vaginal delivery or pregnancy termination beyond 12 weeks gestation (as patulous cervical os may affect VAS score).
* Any previous deliveries had been by cesarean section.
* Immediately postmenstrual or 1 week after pregnancy termination.
* They were willing to complete the study questionnaires.
* All women had to be alert, oriented, and cooperative to respond easily to VAS.

Exclusion criteria were:

* Current pregnancy.
* Prior vaginal delivery.
* History of cervical stenosis.
* Current pelvic inflammatory disease.
* Uterine anomalies.
* Undiagnosed abnormal uterine bleeding.
* Fibroids distorting the uterine cavity.
* Patients using chronic NSAIDs or on chronic pain medication. We randomized participants in a 1:1 ratio to cough and control groups. A statistician not directly involved in the study prepared a computer generated randomization list and placed the allocation information in sequentially numbered sealed envelopes that were opened according to the attendance of the subjects after signing the informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
The level of pain experienced at different steps of IUD insertion measured by a visual analogue scale (VAS). | Up to 22 months
  The primary outcome measure was the level of pain experienced at different steps of IUD insertion measured by a visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Elkhouly, MD, Principal Investigator — Assistant professor of obstetrics and gynecology, faculty of medicine menoufia university
Locations (1):
- Menoufia university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No